CLINICAL TRIAL: NCT07216690
Title: Pregnenolone as a Treatment for Cannabis Intoxication
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00526530; R21DA063854 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Intoxication
Keywords: cannabis; pregenolone; cannabis intoxication; THC; delta-9-thc; CB1 receptor
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol; Pregnenolone

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, within subjects
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind, double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo Brownie and Capsules (Placebo Comparator): Placebo brownie, 0mg THC; two 0 mg pregnenolone capsules
  Interventions: Drug: Placebo; Drug: Placebo brownie
- Cannabis/THC brownie and Placebo Capsules (Placebo Comparator): 25mg Cannabis/THC Brownie; two 0 mg pregnenolone capsules
  Interventions: Drug: Cannabis; Drug: Placebo
- Cannabis/THC Brownie and Pregnenolone, low dose (Experimental): 25mg Cannabis/THC Brownie; one 250 mg pregnenolone capsule and one 0 mg pregnenolone capsule
  Interventions: Drug: Cannabis; Drug: Pregnenolone 250 mg
- Cannabis/THC Brownie and Pregnenolone, high dose (Experimental): 25mg Cannabis/THC Brownie and two 250 mg pregnenolone capsules
  Interventions: Drug: Cannabis; Drug: Pregnenolone 500 mg

INTERVENTIONS:
Drug: Cannabis — Cannabis brownie, 25mg THC
  Other Names: delta-9-tetrahydrocannabinol; THC; delta-9-THC
  Arms: Cannabis/THC Brownie and Pregnenolone, high dose; Cannabis/THC Brownie and Pregnenolone, low dose; Cannabis/THC brownie and Placebo Capsules
Drug: Pregnenolone 250 mg — Pregnenolone, low dose, one 250mg pregnenolone capsule and one 0 mg pregnenolone capsule
  Other Names: Pregnenolone
  Arms: Cannabis/THC Brownie and Pregnenolone, low dose
Drug: Pregnenolone 500 mg — Pregnenolone, high dose, two 250 mg pregnenolone capsules
  Other Names: Pregnenolone
  Arms: Cannabis/THC Brownie and Pregnenolone, high dose
Drug: Placebo — Placebo capsule, 0mg
  Arms: Cannabis/THC brownie and Placebo Capsules; Placebo Brownie and Capsules
Drug: Placebo brownie — Placebo brownie, 0mg THC
  Arms: Placebo Brownie and Capsules

SUMMARY:
The present study will characterize the ability of pregnenolone to reverse the acute intoxication and associated symptoms of cannabis. Healthy adults with a history of cannabis use will be recruited to participate in a placebo-controlled, within-subject crossover study at Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). By clarifying the ability of pregnenolone to reverse cannabis intoxication symptoms, this study will pave the way for larger clinical studies that provide a foundation for the development of future CB1-receptor NAM medications that could be applied in emergency situations and potentially validate pregnenolone as a treatment for cannabis intoxication.

DETAILED DESCRIPTION:
This human laboratory study will characterize the ability of pregnenolone to reverse the acute cannabis intoxication using measures of subjective drug effects, cardiovascular responses, and cognitive performance. Participants (n=16) will complete four double-blind, randomized, outpatient sessions. In each session, participants will self-administer cannabis containing either 0 mg THC (placebo) or 25 mg THC (active) via an oral route of administration. Ninety minutes after cannabis administration, participants will self-administer two oral capsules containing either 0 mg pregnenolone or 250 mg pregnenolone for a total of either 0 mg, 250 mg, or 500mg pregnenolone. Assessments will include subjective drug effect instruments, a battery of cognitive and psychomotor performance tasks, and physiological measures. Sessions will be conducted at a target rate of once per week. Results from this study of pregnenolone could have far-reaching clinical implications: not only would results provide conceptual support for NAMs as treatments for cannabis intoxication but may posit pregnenolone itself as a novel pharmacotherapeutic that could reduce the burden of ineffective and potentially harmful medications currently used in the treatment of cannabis intoxication in emergency settings. If pregnenolone is shown to be effective, additional drug development can be done to determine the best formulation, dose, and route of administration for maximal clinical benefit. Should pregnenolone not reverse THC intoxication completely, development of analogs with greater efficacy can be explored.

ELIGIBILITY:
Inclusion Criteria

* Ages 18-65
* Good general health based on screening procedures (e.g. physical exam, blood testing, psychiatric evaluation)
* Systolic blood pressure <140 mm Hg, diastolic blood pressure < 90 mm Hg, and heart rate <110 bpm at screening and at baseline for dosing session
* Body mass index (BMI) in the range of 18 to 36 kg/m2
* Cannabis use within the past three years but none in the month prior to the first test session
* Negative urine test for illicit substance use and negative breath alcohol test (0% breath alcohol concentration) at screening and before study sessions

Exclusion Criteria

* Use of psychoactive substances (aside from nicotine, caffeine, and alcohol) in the month prior to study initiation
* Current use of over the counter (OTC) drugs, supplements/vitamins, or prescription medications that, in the opinion of the investigator or medical staff, will impact the participant's safety.
* Current use of any prescription or non-prescription medications, including herbal medicines and supplements, that are known to interact with cannabis or pregnenolone
* Self-report or ECG indicating clinically significant cardiovascular conditions, including coronary artery disease, stroke, angina, uncontrolled hypertension, arrhythmias (e.g. atrial fibrillation), heart valve placement, or TIA in the past year.
* History of hormone-sensitive conditions, including but not limited to gynecologic cancers (breast, ovarian, uterine, etc), endometriosis, uterine fibroids, thyroid, pituitary and/or adrenal syndromes, polycystic ovarian syndrome, etc.
* Epilepsy or a history of seizures
* Any of the following laboratory values during screening or upon admission:

  * AST > 165 U/L (normal range 19-55)
  * ALT > 216 U/L (normal range 19-72)
  * Alkaline phosphatase > 1.5x upper limit of normal (ULN)
  * Total bilirubin >1.5 ULN
  * Glomerular filtration rate (EGFR) < 60 ml/min/1.73m2
* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders, or bipolar I or II disorder
* Other unstable and/or compromising medical or psychiatric conditions based on clinical interview and/or MINI results that would interfere with participant safety as determined by study physician, including suicidal ideation and/or attempt, psychosis
* Previous diagnosis and treatment for Cannabis Use Disorder
* Urine drug screen (e.g. Healgen Scientific 14 Panel Rapid Drug Test) indicating the presence of substances including amphetamines, barbiturates, benzodiazepines, cocaine, opioids (including fentanyl), PCP, and THC at screening and prior to study sessions
* Breathalyzer screen indicating presence of alcohol at screening and prior to study sessions
* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing
* Women who are of childbearing potential and sexually active who are not practicing an effective means of birth control including oral contraceptives, progestin implant, transdermal birth control patch, intrauterine device (IUD) or vaginal ring. Women who report use of condoms or diaphragm must use a "double-barrier" method of contraception (i.e. diaphragm and condoms).
* SBP >/= 140, DBP >/= 90, or pulse >/=100 during screening and/or prior to dosing session
* Has donated blood within 30 days of the study
* Allergy to eggs or other food allergies that would make ingestion of brownie mix unsafe.
* Use of concomitant medications, including herbal medicines and botanical supplements, that are strong inhibitors or inducers of CYP3A4 and CYP2C9

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean Peak Change From Baseline Drug Effect as Assessed by the Drug Effect Questionnaire (DEQ) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline rating (0-100) of Drug Effect items related to stimulation (e.g., alertness) and sedation (e.g., sleepy/tired) on the DEQ, a visual analog scale (VAS) self-report questionnaire, with 0 being no effect and 100 being maximum effect.
Mean peak change from baseline psychomotor performance as assessed by the Digit Symbol Substitution Task (DSST) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Mean peak change from baseline total correct trials in 90-seconds. Minimum score of 0 but no maximum score (higher scores indicate better performance).
Mean peak change from baseline working memory performance as assessed by the Paced Auditory Serial Addition Task (PASAT) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Computerized version of Paced Auditory Serial Addition Task administered to assess working memory performance. Mean peak change from baseline total correct trials out of 90 recorded is primary outcome (higher scores indicate better performance).
Mean Peak Levels of Blood Pregnenolone, THC, and THC metabolites (11-OH-THC, and THCCOOH. ) | baseline and 1.5, 2, 3, 4, and 6 hours post-dosing
  Mean peak levels of pregnenolone, THC, and the THC metabolites 11-OH-THC, and THCCOOH in the blood of participants.
Mean Peak Change from Baseline Psychotomimetic effects as assessed by the Psychotomimetic States Inventory (PSI) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline rating of PSI, a 48-item scale designed to measure psychotomimetic effects resulting from psychoactive substance use. Participants rate each item on a four-point visual analog scale, 0 (not at all), 1 (slightly), 2 (moderately), or 3 (strongly). Higher score worse effects.
Mean Peak Change From Baseline Heart Rate | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline heart rate (as measured by beats per minute)
Mean Peak Change From Baseline Blood Pressure (mmHg) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline blood pressure (systolic and diastolic)

SECONDARY OUTCOMES:
Mean peak change from baseline psychomotor performance (attempted and percentage correct) as assessed by the Digit Symbol Substitution Task (DSST) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Mean peak change from baseline total number attempted and percentage correct trials in 90-seconds. Minimum score of 0 but no maximum score (higher scores indicate better performance).
Mean peak change from baseline working memory performance (reaction time) as assessed by the Paced Auditory Serial Addition Task (PASAT) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Computerized version of Paced Auditory Serial Addition Task administered to assess working memory performance. Mean peak change from baseline reaction time on correct trials out of 90 recorded is secondary outcome (faster reaction times indicate better performance).
Mean Peak Change From Baseline Drug Effect (positive effect) as Assessed by the Drug Effect Questionnaire (DEQ) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline rating (0-100) of "positive" Drug Effect items (e.g., "like"; "want more) on the DEQ, a visual analog scale (VAS) self-report questionnaire, with 0 being no effect and 100 being maximum effect.
Mean Peak Change From Baseline Drug Effect (negative effect) as Assessed by the Drug Effect Questionnaire (DEQ) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline rating (0-100) of negative Drug Effect items (e.g., "dislike") on the DEQ, a visual analog scale (VAS) self-report questionnaire, with 0 being no effect and 100 being maximum effect.
Mean Peak Change From Baseline Drug Effect (cannabis specific) as Assessed by the Drug Effect Questionnaire (DEQ) | baseline and 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dosing
  Mean Peak change from baseline rating (0-100) of cannabis-specific Drug Effect items (e.g., "paranoid"; "munchies") on the DEQ, a visual analog scale (VAS) self-report questionnaire, with 0 being no effect and 100 being maximum effect.
Mean Peak Changes from Baseline in ratios of blood pregnenolone levels to blood levels of THC and 11-OH-THC | baseline and 1.5, 2, 3, 4, and 6 hours post-dosing
  Peak blood levels of pregnenolone will be compared to peak blood levels of THC and 11-OH-THC across the timepoints throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Wolinsky, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States